CLINICAL TRIAL: NCT03754920
Title: The Physical and Mental Effects of Prolonged Fasting With Meditation and Mild Physical Exercise
Brief Title: Prolonged Fasting With Meditation and Mild Physical Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ShanghaiUTCMjialijun
Record Dates: First submitted 2018-11-14; First posted 2018-11-27 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-10

CONDITIONS: Fasting
Keywords: prolonged fasting; meditation; physical exercise
MeSH Terms: conditions — Fasting; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prolonged fasting (Experimental): Participants fast for five days, without any food, except unlimited mineral water, and do some fitness regimen(such as meditation and mild physical exercise ).
  Interventions: Behavioral: prolonged fasting

INTERVENTIONS:
Behavioral: prolonged fasting — Fasting for 5 days: Fasting with some fitness regimen, such as meditation and mild physical exercise;
  Feeding for 3 days: Gradually distribute participants with rice flour, porridge and juice.

SUMMARY:
To determine the feasibility, safety and efficacy of fasting, participants are recruited in a 5-days fasting ( without any food, except unlimited mineral water),and do some fitness regimen (such as meditation and mild physical exercise ) during fasting.The samples will be collected from participates and subjected to comprehensive analysis ,including routine medical examination in blood, metabonomics and proteomics anlysis in serum and urine samples, gut microbiome analysis in stood samples, and so on.

DETAILED DESCRIPTION:
1. Recruiting: 45 healthy people will be included in the clinical trial according to the Inclusion criteria and exclusion criteria.
2. Fasting : Participants fast for five days, without any food, except unlimited mineral water. Participants will do some fitness regimen (such as meditation and mild physical exercise ) during fasting.
3. Re-feeding: Gradually distribute participants with rice flour, porridge and juice in the next 3 days.
4. Follow-up :The health checklist is similar with that during fasting on the first month.
5. Data processing, statistics and analysis. Diet monitoring: The intake of glucose decreases, while the burning of fat increases, which can down-regulate glucose level in blood, up-regulate ketone level in urine. Thus, the fasting situation of participants can be monitored by the variation of blood glucose and urine ketone.

ELIGIBILITY:
Inclusion criteria

1. 18-65 years old, no nationality limitation, no gender limitation;
2. Male weight ≥ 50 kg, female weight ≥ 45 kg；BMI: 19-28 kg/m²;
3. The index of physical examination is in line with health standards;
4. People who have gone through a 7-day fasting before ;
5. Agree to take part in the trials and sign the informed consent form.

Exclusion criteria

1. People with unhealthy habits, such as smoking(5 cigarettes per day, or can not stop smoking in the trial), excessive drinking(drink regularly in the recent 6 months or more than 14 units of alcohol per week (1 unit = 360 ml beer or 45 ml alcohol with 40% spirits or 150 ml wine)) ;
2. People who processed fasting within one month;
3. Pregnancy, current breast-feeding or menstrual period;
4. People who are marantic, malnourished or anorectic;
5. People who have cardiovascular disease(coronary heart disease, atherosclerosis, arrhythmia, etc), serious metabolic and psychiatric disorders(hypertension, type 2 diabetes, hyperthyroidism, etc.);
6. People who have Mental illness, cancer, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), syphilis, human immunodeficiency virus (HIV) antibody positive.
7. people who has mental disorders according to the scales(Hamilton Anxiety Scale、Self-Rating Anxiety Scale、Self-rating depression scale)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-04-09 (Estimated); Study Completion 2019-09-09 (Estimated)

PRIMARY OUTCOMES:
Weight | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Changes in weight will be assessed.
Blood glucose | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Changes in blood glucose will be assessed.
Insulin | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in insulin will be assessed.
Blood pressure | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Changes in blood pressure will be assessed.
Waistline | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Changes in waistline will be assessed .
IGF-1 | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in IGF-1 will be assessed.
Pulse Rate | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Changes in pulse rate will be assessed.
Blood lipid test | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in blood including HDL, LDL, TG, CHO and ect. will be assessed.
Urine test | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in urine including uric acid and ect. will be assessed.
Liver and renal function test | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in liver and renal function including AST,ALT,ALP, TP,ALB, Urea, Crea and ect will be assessed at 7：30 am.
Serum metabolomics analysis | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Serum samples were collected and serum metabolomics (carbohydrate, lipid, amino acid and ect.) were sequenced and analyzed by High-throughput sequencing.

SECONDARY OUTCOMES:
Urinary ketone | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Changes in urinary ketone will be assessed.
Vitamin examination | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in vitamin including vitamin C,D,E and etc. will be assessed.
Thyroid function | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in Thyroid function test including FT3，FT4，TSH will be assessed.
Inflammatory factors | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Changes in inflammatory factors includingIL1, IL2, IL6, IL10，TNF ,TGFβ and etc. will be assessed.
Gut microbiome | Day 0, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8; 1 month and 3 months post fasting
  Stool samples were collected in time if possible and analyzed the composition /function of the intestinal microflora by High-throughput sequencing
Self-rating depression scale； | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  The Scale ,includes half of items ues positive words and half is negatively,which could assess symptoms of depression. Item responses are ranked from 1 to 4, and higher scores correspond to more frequent symptoms. For each item,patients give a score according to whether the item has occurred: 1 = never/very rarely; 2 = once in a while/some of the time/occasionally; 3 = relatively often/very often/often; 4 = most of the time/always. Each items points accumulated as raw scores,the lowest raw score is 20 points, the highest raw score is 80 points. The raw scores multiply by 1.25, taking the integer part as the standard scores.The scale standard scores were used to define four categories of depression severity: within normal range or no significant psychopathology (below 51points); presence of minimal to mild depression (51-60points); presence of moderate to marked depression (61-70points).
Self-Rating Anxiety Scale； | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  The Scale contains 20 questions. Each question is scored on a scale of 1-4 (never, some of the time, relatively often, most of the time). There are fifteen questions involved in the assessment could indicate the increase of anxiety levels, and rest of the questions assessment would decrease of the anxiety levels.Each items points accumulated as raw scores,the lowest raw score is 20 points, the highest raw score is 80 points. The raw scores multiply by 1.25, taking the integer part as the standard scores.The scale standard scores were used to define four categories of anxiety severity: within normal ranger no significant psychopathology (25-49points); presence of mild to moderate anxiety levels (50-59points); severe anxiety levels (60-69points); and presence of extreme depression (70-100points).
Hamilton Anxiety Scale | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Symptoms of generalized anxiety disorder as measured by the Hamilton Anxiety Scale (HAM-A) at 1 day、4 day、6 day、9 day、40 day. Each item is scored on a scale from 0 (not present) to 4 (severe) with a total score range of 0-56. Changes in HAM-A scores are calculated as the difference between the baseline HAM-A scores and scores at 1 day、4 day、6 day、9 day、40 day.
Hamilton Depression Scale | Day 0, day 3, day 5, day 8; 1 month and 3 months post fasting
  Remission according to HAM-D: HAM-D17 score less than or equal to (=<) 7 or a HAM-D7 score =< 3. HAM-D17: standardized, clinician-administered rating scale; assesses 17 items characteristically associated with major depression. Individual items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe. Total score: 0 to 66; higher score indicates more depression. HAM-D7: subset of HAM-D17; assesses 7 items associated with major depression. Total score: 0 to 26; higher score indicates more depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Jia, Ph.D., Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided